CLINICAL TRIAL: NCT02725502
Title: Effect of Linagliptin on Incretin Axis in Type 1 Diabetes
Brief Title: Incretin Axis in Type 1 Diabetes Mellitus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Sanjay K. Bhadada, Associate Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Type 1 Diabetes Mellitus
Record Dates: First submitted 2014-01-20; First posted 2016-04-01 (Estimated); Last update posted 2016-04-01 (Estimated); Status verified 2016-03

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: T1DM; Linagliptin; mix meal test
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Linagliptin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Linagliptin treatment group (Active Comparator): Group will receive linagliptin ( 5 mg / day ) for 3 months in addition to their insulin
  Interventions: Drug: Linagliptin
- Placebo group (Placebo Comparator): Group will receive placebo for 3 months in addition to their insulin
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Linagliptin — Baseline HbA1C will be assessed. Before starting treatment with linagliptin or placebo Mixed meal test will be conducted with the standard protocol. Morning dose of insulin to be omitted on the day of mixed meal test. During the mixed meal test glucose, C-peptide, GLP1 and glucagon will be measured at 0, 30, 60, 120, 180 minutes. 72 hour blood glucose profile to be monitored with continuous glucose monitoring system (CGMS). Markers of glucose control and glucose variability will be measured. Then we will randomly divide these patients in two group (linagliptin and placebo group). After 3 month period 72 hour blood glucose profile, HbA1C and Mixed meal test will be repeated to document any change in blood glucose profile.
  Arms: Linagliptin treatment group
Drug: Placebo — Baseline HbA1C will be assessed. Before starting treatment with linagliptin or placebo. Mixed meal test will be conducted with the standard protocol. Morning dose of insulin to be omitted on the day of mixed meal test. During the mixed meal test glucose, C-peptide, GLP-1 and glucagon will be measured at 0, 30, 60, 120, 180 minutes. 72 hour blood glucose profile to be monitored with CGMS. Markers of glucose control and glucose variability will be measured. Then we will randomly divide these patients in two group (linagliptin and placebo group). After 3 month period 72 hour blood glucose profile, HbA1C and Mixed meal test will be repeated to document any change in blood glucose profile.
  Arms: Placebo group

SUMMARY:
Type 1 diabetes is an autoimmune disorder characterized by beta cell destruction resulting in insulinopenia. Currently it is being treated with insulin. Dipeptidylpeptidase inhibitors (DPP4 inhibitors e.g. linagliptin & sitagliptin) has been used for type 2 diabetes mellitus (T2DM) traditionally. Previous studies has shown that it is also effective in type 1 diabetes mellitus (T1DM), but the mechanism of action not well understood. This study will evaluate possible mechanism of action of linagliptin in T1DM patients.

DETAILED DESCRIPTION:
Glucose is the most important physiologic substance involved in the regulation of insulin release. The effect of glucose on the beta cell is dose related. Dose-dependent increases in concentrations of insulin and C-peptide and in rates of insulin secretion have been observed after oral and intravenous glucose loads with 1.4 units of insulin, on average, being secreted in response to an oral glucose load as small as 12 g. The insulin secretory response is greater with oral compared to intravenous glucose administration. This difference in insulin secretion is known as the incretin effect. This enhanced response to oral glucose has been interpreted as an indication that absorption of glucose by way of the gastrointestinal tract stimulates the release of hormones and other mechanisms that ultimately enhance the sensitivity of the beta cell to glucose. The release of insulin from the beta cell after a meal is facilitated by a number of gastrointestinal peptide hormones, including GIP (Glucose dependent insulinotropic peptide), cholecystokinin, and GLP1 (Glucagon like peptide 1). These hormones are released from small-intestinal endocrine cells postprandialy and travel in the bloodstream to reach the beta cells, where they act through second messengers to increase the sensitivity of these islet cells to glucose. In general, these hormones are not themselves secretagogues, and their effects are evident only in the presence of hyperglycemia. This incretin effect could account for the greater beta-cell response observed after oral as opposed to intravenous glucose administration.

GLP1, the most potent of the incretin peptides, lowers glucose in patients with T2DM by stimulating endogenous insulin secretion and perhaps by inhibiting glucagon secretion and gastric emptying. Treatment with supra physiologic doses of GIP during hyperglycemia has been shown to augment insulin secretion in normal humans but not in individual with diabetes mellitus. Although cholecystokinin has the ability to augment insulin secretion in humans, it is not firmly established whether it is an incretin at physiologic levels. Its effects are also seen largely at pharmacological doses.

Type 1 diabetes (T1DM) is characterized by autoimmune pancreatic β cell destruction and insulin deficiency resulting in hyperglycemia. Insulin is the mainstay of treatment in T1DM. There are few study which showed effectiveness of OHA (oral hypoglycemic agents) in T1DM.

Linagliptin is a dipeptidyl peptidase 4 (DPP4) inhibitor. It increases endogenous glucagon like peptide 1 levels by inhibiting its rapid metabolism through the dipeptidyl peptidase 4 enzyme. It is currently Food and Drug Administration (FDA) approved for the treatment of Type 2 diabetes (T2DM ) as mono therapy or in combination with insulin or other oral hypoglycemic agents. Increasing endogenous glucagon like peptide 1 levels in patients with T2DM has been shown to significantly improve postprandial glucose levels by both increasing glucose-dependent insulin release and reducing glucagon levels.

Studies had shown that sitagliptin, a DPP4 inhibitor is effective in T1DM. But the mechanism of action is unknown. In this study the investigators want to investigate the effect of linagliptin, another DPP4 inhibitor on the glycaemic profile, HbA1C and glycaemic variability in patients with T1DM. The investigators also will assess the GLP1 and glucagon response during mixed meal test to identify the potential mechanism of this novel form of therapy. These out come parameters will be compared with placebo treated T1DM patients. During this study patients will be monitored for any adverse effect like nausea, vomiting, pancreatitis. Serum urea, creatinin, amylase and lipase will be monitored monthly.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adult, aged 15 to 30 years
* Duration of type 1 Diabetes Mellitus for 6 months or more, as established by medical history
* Current treatment with multiple injections of insulin for at least 3 months prior to screening visit; and using the same insulin during the last 1 month
* HbA1c < 8%
* Body mass index (BMI) < 25 kg/mt2
* Euthyroid patient. If thyroid dysfunction is present then thyroid function test (TFT) should be normal at the time of study ( with medication)

Exclusion Criteria:

* On pramlintide, metformin, GLP1 agonist or DPP4 inhibitor. If taking this drugs then stop them 2 wk prior to study.
* On prokinetics & proton pump inhibitor (PPI). If taking this drugs then stop them 2 wk prior to study
* Creatinine of >1.5 mg/dl or a calculated creatinin clearance of <50 ml/min or overt proteinuria.
* Fasting blood glucose (FBG) < 72 or > 180 in the day of mixed meal test (MMT)
* Pregnant
* Seriously ill patients
* Presence of gastroparesis ( if history is suggestive of autonomic neuropathy or gastroparesis then gastric emptying study to be done to rule it out)
* Type 1 Diabetes Mellitus for less than 6 months duration
* Presence of celiac disease

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-07; Primary Completion 2016-04 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Effect of Linagliptin on HbA1c in T1DM patients | After 3 months of the starting of the treatment
  Change in HbA1C in linagliptin group as compared to placebo group
Effect of Linagliptin on glycemic variability in T1DM patients | After 3 months of the starting of the treatment
  Change in glycemic variability (CGMS indices) in linagliptin group as compared to placebo group
Effect of Linagliptin on insulin requirement in T1DM patients | After 3 months of the starting of the treatment
  Change in insulin requirement in linagliptin group as compared to placebo group

SECONDARY OUTCOMES:
Effect of linagliptin on GLP1 level during mixed meal test in T1DM patients | after 3 months of the starting of the treatment
  Change in Area under the curve (AUC) of GLP1 during mixed meal test in linagliptin group as compared to placebo group
Effect of linagliptin on glucagon level during mixed meal test in T1DM patients | after 3 months of the starting of the treatment
  Change in Area under the curve (AUC) of glucagon during mixed meal test in linagliptin group as compared to placebo group

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Kr Bhadada, MD, DM, Principal Investigator — Department of Endocrinology, PGIMER, Chnadigarh India
Locations (1):
- Department of Endocrinology, PGIMER, Chandigarh, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No